CLINICAL TRIAL: NCT03766802
Title: Effects of Wearable Technology and Smart Mobile Phone Applications Based Exercise Training and Supervised Exercise Training in Patients With Type 2 Diabetes
Brief Title: Effects of Wearable Technology and Smart Phone Applications Based Exercise Training in Patients With Type 2 Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 09.2017.604
Record Dates: First submitted 2018-12-01; First posted 2018-12-06 (Actual); Last update posted 2019-02-01 (Actual); Status verified 2019-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2; Physical activity; exercise behavior; exercise; smart phone; wearable technology; self-management; glycated hemoglobin (HbA1c)
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: Group 1: Wearable watch training group. 3 orientation session Watch notifies 3/week for exercise
  Benefits of watch:
  BP and movement sensors allow to validate if the patient has exercised. Videos for exercises. Trackable and notifiable if patients don't exercise. Group 2: Mobile application training group. 3 orientation session App notifies 3/week for exercise
  Benefits of app:
  Cheaper Trackable and notifiable if patients don't exercise. Group 3: Supervised exercise training in a fitness center for people with DM.
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wearable watch training group. (Active Comparator): Aerobic exercises Strengthening exercises Stretching exercises Balance exercises Dose was increased as person is able to tolerate. Form:intervention is trackable and notifiable if patients don't exercise with smartwatch.
  Frequency:3/week Duration:12 weeks Dosage:Dose was increased as person is able to tolerate.
  Interventions: Behavioral: Wearable watch training group.
- Mobile application training group. (Active Comparator): Aerobic exercises Strengthening exercises Stretching exercises
  Balance exercises Form:intervention is trackable and notifiable if patients don't exercise with smartphone Dose was increased as person is able to tolerate. Frequency:3/week Duration:12 weeks Dosage:Dose was increased as person is able to tolerate.
  Interventions: Behavioral: Mobile application training group.
- Supervised exercise training group (Sham Comparator): Aerobic exercises Strengthening exercises Stretching exercises supervised by a physical therapist
  Interventions: Behavioral: Supervised exercise training group

INTERVENTIONS:
Behavioral: Wearable watch training group. — 3 orientation session Watch notifies 3/week for exercise
  Arms: Wearable watch training group.
Behavioral: Mobile application training group. — 3 orientation session App notifies 3/week for exercise
  Benefits of app:
  Cheaper Trackable and notifiable if patients don't exercise.
  Arms: Mobile application training group.
Behavioral: Supervised exercise training group — 3/week training supervised by a physical therapist
  Arms: Supervised exercise training group

SUMMARY:
The purpose of this study is to estimate the extent to which supported exercise training through wearable technology and mobile application affects glycemic control in comparison to supervised exercise training in patients with Type-2 Diabetes.

DETAILED DESCRIPTION:
The purpose of this study is to estimate the extent to which supported exercise training through wearable technology and mobile application affects glycemic control in comparison to supervised exercise training in patients with Type-2 Diabetes.

Inclusion Criteria:

* Age 18-65
* No other chronic condition
* No exercise training background Block Randomization according to age and sex.

Confirmatory Outcome

- Glycated Hemoglobin (HbA1c)

Explanatory outcomes

* Flexibility
* Level of Physical Activity - IPaQ (METS) and accelerometer
* Hamstring / Quad strength - isokinetic
* Grip strength
* Respiratory function test - F1, FVC, F25, F75, F100
* 6MWT
* Balance - static, dynamic, proprioception, sit-to-stand balance
* Body Muscle Percentage - bioelectrical impedance analysis

ELIGIBILITY:
Inclusion Criteria:

Age 18-65 No other chronic condition No exercise training background

Exclusion Criteria:

* Exclusion criteria are a set of predefined condition that is used to identify subjects who will not be included or who will have to withdraw from a research study after being included.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2018-09-22 (Actual); Study Completion 2019-05-05 (Estimated)

PRIMARY OUTCOMES:
Glycated Hemoglobin (HbA1c) | 5 minutes
  It used as a diagnostic test for diabetes and as assessment test for glycemic control in people with diabetes. It comes in unit of percentage identifies how much glucose is carried on a certain amount of blood. We included people who have 6.5% or more which is the cut point for The International Diabetes Federation and the American College of Endocrinology.

SECONDARY OUTCOMES:
Six-Minute Walk Test | 6 min
  The 6-min walk test (6 MWT) is a submaximal exercise test that entails measurement of distance walked over a span of 6 minutes
The forced vital capacity | 10 minutes
  The forced vital capacity (FVC) is a measurement of the maximum volume of gas a patient can exhale as forcefully and quickly as possible after a maximal inspiration.Pulmonary function test used to determine forced vital capacity. Breathing multiple times into a spirometry, with regular and maximal effort, through a tube that is connected to a computer. The unit for this test is in volume (L). And it will be analyzed as a continuous variable.
Forced expiratory volume | 10 minutes
  Forced expiratory volume (FEV) measures how much air a patient can exhale during a forced breath. Pulmonary function test used to determine Forced expiratory volume.The amount of air exhaled is measured during the first (FEV1), second (FEV2), and/or third seconds (FEV3) of the forced breath. The unit for this test is in volume (L). And it will be analyzed as a continuous variable.
Assessment of muscle strength with isokinetic device | 15 minutes
  An assessment of muscle strength is typically performed as part of a patient's objective assessment.
International physical activity questionnaire short form (IPAQ) | 7 days
  The International Physical Activity Questionnaire (IPAQ) is used as a comparable and standardised self-report measure of habitual physical activity.
Accelerometer | 7 days
  Accelerometer is a device that measures hours of physical activity in a week. The device was placed on the belt of the participants and was collected back after 7 days. Accelerometer collects data on the three-dimensional angles, which explains the direction, frequency, and magnitude of the movement. Total number of hours of physical activity is used to measure whether participants meet the optimal activity level recommended by physical activity guidelines.

OTHER OUTCOMES:
Exercise Adherence Rating Scale (EARS) | 5 minutes
  The EARS enables the measurement of adherence to prescribed home exercise. This may facilitate the evaluation of interventions promoting self-management for both the prevention and treatment of chronic conditions.
Behavioural Regulations in Exercise Questionnaire | 5 minutes
  The Behavioural Regulation In Exercise Questionnaire (BREQ) and its subsequent modifications have become the most widely used measures of the continuum of behavioural regulation in exercise psychology research
HDL / LDL | 5 minutes
  The main goal is to lower LDL-cholesterol and increase HDL-cholesterol. Therefore, HDL and LDL were measured before and after the intervention to identify whether our program had an effect on the cholesterol level. The unit is mmol/L and it comes as a continuous variable.
Triglyceride | 5 minutes
  Triglycerides are a type of fat (lipid) found in people' blood. It was also measured to estimate the extent to which our intervention had effect on the blood-fat level. The unit is mmol/L and it comes as a continuous variable.

CONTACTS AND LOCATIONS:
Overall Officials: Eren Timurtas, PT, MSc, Principal Investigator — Marmara University
Locations (1):
- Faculty of Health Sciences, Istanbul, Maltepe, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.